CLINICAL TRIAL: NCT00839410
Title: Multicentric Cohort of Melanoma Patients in Ile de France Area
Acronym: Melan-Cohort
Status: Completed | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: P020927
Record Dates: First submitted 2009-02-06; First posted 2009-02-09 (Estimated); Last update posted 2019-10-04 (Actual); Status verified 2019-09

CONDITIONS: Melanoma; Genetic Polymorphism
Keywords: skin cancer; melanoma; sentinel lymph node biopsy; bio bank; genetic polymorphism; prospective cohort; cohort; sentinel lymph nodes; tissue samples
MeSH Terms: conditions — Melanoma; Skin Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — DNA,RNA,SERUM,PLASMA,PROTEOMICS
Oversight: Data Monitoring Committee: Yes

SUMMARY:
This is a multicentric prospective cohort of all stage melanoma patients from AP-HP ,the largest consortium of University hospitals over Europe. 7 investigation sites (7 dermatological services of AP-HP) in Ile de France region are involved. 1300 patients will be enrolled and be followed during 10 years.

DETAILED DESCRIPTION:
Melan-Cohort should constitute the first multicentric cohort with various objectives: prognostic, therapeutic, cognitive and medico-economical studies on melanoma. Patients will be recruited in all of the dermatology departments of APHP (dermatology departments from AMBROISE PARE, Saint-Louis, BICHAT-Claude Bernard,Henri-Mondor, Cochin-Tarnier, and Tenon hospitals). For all included patients, a standard file is filled comprising all anatomy-clinical useful data and epidemiologic ones, including sun exposures. Blood is harvested to collect DNA, RNA, serum, plasma at inclusion and at regular intervals and in case of progressive disease. Procedures for sentinel lymph node biopsies have been homogenized. An informed consent is obtained for each patient included in the cohort. A steering committee meets on a regular basis, and genetics or pathology subgroups have been constituted. An electronic CRF is available using the Intranet of APHP hospitals. Specimens are stored using high quality standards.

ELIGIBILITY:
Inclusion criteria :

* age ≥ 18 years
* an informed consent is obtained
* patients with anatomy-pathologically proved melanoma
* the tissue sample of melanoma is available
* the primary melanoma is treated according to the international standard
* absence of a progressive non neoplastic pathology involving life-threatening
* patient living in Ile de France region.
* time limit to entry in the cohort must be:
* within 3 months after Surgical resumption of primary melanoma;
* within 3 months after curative surgical treatment;
* with one month after diagnosis of a transit metastasis or a distant metastasis.

Exclusion criteria :

* refusal of the patient
* pathology sample isn't available
* primary melanoma not being treated according to the international standard
* patient living too far to follow regular visits
* patient diagnosed with a progressive non neoplastic pathology involving life-threatening
* too late to entry and lack of useful stored specimens to research.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults with anatomo-pathologically proved melanoma
Sampling Method: Non-Probability Sample
Enrollment: 1255 (Actual)
Dates: Start 2003-09 (Actual); Primary Completion 2019-10 (Actual); Study Completion 2019-10 (Actual)

PRIMARY OUTCOMES:
Overall survival (0-10 years) Disease free survival (0-10 years) | 10 years

SECONDARY OUTCOMES:
Invasion of sentinel lymph node biopsy | 2003-2009

CONTACTS AND LOCATIONS:
Overall Officials: Philippe Saiag, MD, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Pr Philippe Saiag, Boulogne-Billancourt, Île-de-France Region, France